CLINICAL TRIAL: NCT07234227
Title: Genitourinary Study of Fostering Lactobacillus to Optimize the Microbiome in Women's Health (GUD-FLORA)
Acronym: GUD-FLORA
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00118524
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Recurrent UTIs
Keywords: Recurrent UTI; Microbiome; Probiotic; Vaginal probiotic; Lactobacillus; Urinary tract infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Probiotic Group (Experimental): All patients will receive vaginal probiotic product
  Interventions: Drug: Lactobacillus crispatus probiotic

INTERVENTIONS:
Drug: Lactobacillus crispatus probiotic — Probiotic arm (all patients)
  Other Names: Probiotic; VS-01(TM)

SUMMARY:
The objective of this study is to evaluate the use of a vaginal probiotic in patients with recurrent urinary tract infections (UTIs). Specifically, this study aims to evaluate factors associated with successful colonization with Lactobacillus crispatus - a known "healthy" and protective bacteria in both the vaginal and urinary microenvironments. The study will recruit patients over age 18 with a clinical diagnosis of recurrent UTIs, and will utilize a commercially available Lactobacillus vaginal probiotic. Participants will use the probiotic product with the commercially approved packaging and regimen for a total of 3 months. Vaginal and urinary samples will be obtained at four different timepoints. Participants will also be asked to complete surveys regarding tolerability and acceptability of the probiotic product. Patient samples will be analyzed in the laboratory to understand the effects of the probiotic on the local microbiome. Survey data and demographic information will be housed within the Research Electronic Data Capture (RedCap) secure server. For our primary analysis, Lactobacillus crispatus (L. crispatus) abundance will be measured and used as the outcome variable in a linear regression model evaluating the impact of baseline patient and microbiome characteristics on L. crispatus colonization.

DETAILED DESCRIPTION:
This is a prospective, observational study in patients with recurrent UTIs seeking care in the Duke Division of Urogynecology.

After obtaining informed consent, baseline samples and questionnaires will be completed during an in person visit. Clinical data will be abstracted from the medical record. At the baseline visit, participants will be supplied a 3-month course of the VS-01TM vaginal probiotic, manufactured by Seed Health, Inc. VS-01TM is a commercially available dissolving tablet containing three strains of L. crispatus. The tablet is self-administered vaginally via a supplied applicator.

Participants will follow the recommended dosing regimen (e.g., Days 1, 4, 7, 14, 21, 28, then every other week) to total 3 months.

No existing patient therapies for recurrent UTIs will be discontinued or prohibited during the study period. Patients will be encouraged to continue any stable/existing medications for UTI prevention such as vaginal estrogen. No placebo control will be utilized.

Participants will be supplied with at-home sampling kits for sample collection. Final sampling occurs once month after completion of the probiotic regimen, with samples banked for future analyses to determine whether colonization persists after cessation of the probiotic. Sampling will occur at baseline and at weeks 4, 10, and 16. Each sampling time point will include a urine sample and a vaginal swab. The baseline sample will also include a pH test via pH paper strip.

Home sampling procedures will be similar to those recently published by a large consortium. Participants will return sampling kits via pre-paid, pre-addressed shippers through our laboratory account. Due to the at-home nature of patient sample collection, no additional visits to clinic will be required. Patients will have access to routine clinic visits per standard of care.

Upon receipt in the lab, samples will be processed, and DNA will be extracted. Prepared samples with positive and negative controls will be evaluated for microbial abundance. For our primary analysis, absolute abundance of L. crispatus at baseline and subsequent timepoints will be evaluated using digital droplet PCR. In addition, the investigators will plan to pursue additional funding for sequence-based analyses of L. crispatus and other species. For these additional analyses, samples would be submitted to the Duke Microbiome Core for library preparation, amplification, and sequencing of the full-length 16S rRNA gene. Taxonomic identification will be performed with standard pipelines and relative abundance of L. crispatus and other species will be quantified.

With respect to survey data, all will be completed electronically either in clinic (baseline via iPads), or at home (link sent to designated email), and stored through Research Electronic Data Capture (REDCap). The questionnaires utilized are the Vulvovaginal Symptoms Questionnaire (VSQ) and an acceptability questionnaire. These are validated questionnaires to assess patient tolerability and acceptability, respectively, of the vaginal probiotic regimen.

ELIGIBILITY:
Inclusion Criteria

* English-speaking
* ≥ 18 years of age
* Diagnosed with recurrent urinary tract infections (UTIs). Specifically, participants will have had 3 UTIs over the past 12 months or 2 UTIs over the past 6 months. At least one of these UTIs must be culture-proven. For UTIs to count for this study, if not culture-proven they must involve the onset of UTI-related symptoms (dysuria, urgency, frequency, suprapubic pain, or urinary changes, etc) with prescription of antibiotics directed at UTI treatment.

Exclusion Criteria

* Chronically self-catheterize.
* Currently use of a vaginal pessary.
* Have used a vaginal probiotic in the prior 3 months.
* Are pregnant or within 1 year postpartum.
* Have poorly controlled diabetes with an A1c of 9 or greater.
* Are considered immunocompromised
* Are unable to personally provide legal consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Relative abundance | 10 weeks
  The primary endpoint is relative abundance of vaginal L. crispatus after several months of vaginally inserted L. crispatus probiotics.

SECONDARY OUTCOMES:
Number of participants with Vaginal - Urinary Correlation | Baseline, 4, 10, and 16 weeks
  Correlations in vaginal and urinary L. crispatus, at baseline and several timepoints after initiation and cessation of probiotic.
Tolerability of a vaginal probiotic regimen as measured by the Vulvovaginal Symptoms Questionnaire (VSQ) | Baseline, 4, 10, and 16 weeks
  A higher score on the VSQ (range of 0 to 21) indicates lower tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Nazema Siddiqui, MD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: Yes